CLINICAL TRIAL: NCT04327843
Title: Reducing the Burden of Chronic Psychotic Disorders in Tanzania
Brief Title: Reducing the Burden of Chronic Psychotic Disorders in Tanzania (CAPACITY)
Acronym: CAPACITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor of Psychiatry and of Neurology, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-17-19; R21MH114700 (NIH)
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Medication Nonadherence; Schizo Affective Disorder
Keywords: nonadherence; Schizophrenia; Africa; Schizoaffective
MeSH Terms: conditions — Schizophrenia; Medication Adherence; Psychotic Disorders | interventions — haloperidol decanoate; Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAE + LAI (Experimental): Customized Adherence Enhancement (CAE) + Long-Acting Injectable Antipsychotic (LAI)
  Interventions: Behavioral: Customized Adherence Enhancement; Drug: Haloperidol Decanoate

INTERVENTIONS:
Behavioral: Customized Adherence Enhancement — Customized Adherence Enhancement (CAE): CAE targets key areas relevant to adherence in chronic psychotic disorders (CPD): 1.) inadequate understanding of mental disorder, 2.) lack of adequate medication-taking routines, 3.) poor communication with care providers and 4.) substance use which interferes with adherence and recovery. CAE delivered components are selected based upon findings from the ROMI and AMSQ. CAE will be delivered in approximately 8 sessions by a nurse interventionist, ideally at the same time that the long-acting injectable (LAI) is administered.The intervention is guided by a detailed manual and uses components and resources that are available in lower- and middle-income countries (LMICs). Social worker interventionists will be trained to deliver CAE-L.
  Other Names: CAE
Drug: Haloperidol Decanoate — Long-acting injectable (LAI): Patients on oral haloperidol will be switched to haloperidol decanoate per manufacturer's package insert. Individuals not on antipsychotic medication at the time of screening assessment or who are on a different antipsychotic medication, will receive an oral tolerance test (OTT) consisting of up to 14 days of oral haloperidol 2-5 mg once or twice daily. If the OTT suggests good tolerability, the participant will then receive LAI (haloperidol decanoate) intramuscularly after completion of baseline assessments. Dosing of LAI will be as clinically indicated using conservative dosing to minimize drug-related adverse effects. In the CWRU studies, mean end-point dose of haloperidol decanoate was 68.0 mg, SD 21.1, Range 50-100 mg/monthly injection. It is anticipated that patients will continue on the same dose for 6 months, although dose changes will be permitted based upon clinical status. Each study participant will receive up to 8 injections during the study.
  Other Names: Haldol Decanoate

SUMMARY:
The proposed, three phase project will refine and test a first-ever care approach in SSA that combines LAI with a behavioral program specifically intended to promote medication adherence in chronic psychotic disorders (CPDs). In addition to the novel focus, innovative elements include: 1.) a manualized curriculum that targets specific barriers and facilitators to medication adherence in Tanzanians with CPD, 2.) targeting known, high-risk individuals with CPD (those who miss ≥20% of prescribed antipsychotic medication, and 3.) using existing injection clinic health workers to deliver the adherence promotion program. Strengths include the highly generalizable methods and use of LAIs that are available in low-resource settings.

DETAILED DESCRIPTION:
In this Phase 3 portion, the study team will select appropriate measures, train staff and build capacity in measure implementation, and finalize the intervention for delivery by healthcare workers. Finally, in a training/proof-of-concept exercise, the healthcare workers will implement the adapted CAE-L in a high-risk sample of Tanzanians with CPD (individuals with schizophrenia or schizoaffective disorder who have had recent medication adherence problems). Taken together, the proposed project has substantial public health importance. It will provide the prerequisite materials, training and infrastructure needed for a prospective trial in reducing CPD burden and improving brain health in Tanzania and other countries in Sub-Saharan Africa.

The focus of this project is on feasibility, patient acceptability, and research capacity-building. Therefore a specific hypothesis is not being tested. The investigators will assess descriptive statistics and change from baseline in the primary and secondary measures using standard pre-post techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Diagnosis of schizophrenia or schizoaffective disorder
* Known to have medication treatment adherence problems as identified by the TRQ (20% or more missed medications in past week or past month)
* Ability to be rated on psychiatric rating scales
* Willingness to take long-acting injectable medication
* Able to provide written, informed consent to study participation

Exclusion Criteria:

* History of allergy or intolerance to haloperidol or haloperidol decanoate
* Individuals on long-acting injectable antipsychotic medication immediately prior to study enrollment
* Medical condition or illness, which in the opinion of the research psychiatrist, would interfere with the patient's ability to participate in the trial
* Physical dependence on substances (alcohol or illicit drugs) likely to lead to withdrawal reaction during the course of the study in the clinical opinion of the treated research psychiatrist
* Immediate risk of harm to self or others
* Female who is currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- MUHAS, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mbwambo J, Kaaya S, Lema I, Burant CJ, Magwiza C, Madundo K, Njiro G, Blixen CE, Cassidy KA, Levin JB, Sajatovic M. An interventional pilot of customized adherence enhancement combined with long-acting injectable antipsychotic medication (CAE-L) for poorly adherent patients with chronic psychotic disorder in Tanzania. BMC Psychiatry. 2022 Jan 27;22(1):62. doi: 10.1186/s12888-022-03695-8. PMID 35086504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study setting was Muhimbili National Hospital, a 70-bed national referral hospital located in urban Dar es Salaam, Tanzania.
  Patients were referred from 4 catchment zones that include 3 regional public and private hospitals and were recruited from inpatient and outpatient settings.
  19 adult patients ≥ age 18 with schizophrenia who self-reported missing 20% or more of antipsychotic medication demonstrating poor adherence.
Pre-assignment Details: 38 individuals were assessed for preliminary eligibility. 16 people were excluded, 5 were unable to contact, 2 were not interested, 3 did not meet criteria, and 6 were no-shows for screening.
  22 provided informed consent initially. 2 of these people failed the oral tolerance test and 1 did not complete baseline measures.
  19 participants enrolled and attended visits 1-6 and 18 attended all 7 visits.
Groups:
- CAE + LAI Treatment: The sample comprised adult patients ≥ age 18 with schizophrenia who self-reported missing 20% or more of antipsychotic medication within the last month, an established benchmark for poor adherence who were given a long-acting injectable antipsychotic medication and a customized adherence enhancement behavioral intervention (CAE-L).
Period: Baseline Assessment
Arm/Group | CAE + LAI Treatment
Started | 19
Completed | 19
Not Completed | 0
Period: Week 13 Assessment
Arm/Group | CAE + LAI Treatment
Started | 19
Completed | 19
Not Completed | 0
Period: Week 25 Assessment
Arm/Group | CAE + LAI Treatment
Started | 19
Completed | 18
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.79 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Marital status [Count of Participants; unit: Participants]
  Single/never married | 12
  Married | 2
  Separated/divorced | 4
  Widowed | 1
Educational level [Mean (Standard Deviation); unit: years] | 8.37 (2.99)
Employment [Count of Participants; unit: Participants]
  Full-time | 4
  Part-time | 3
  Unemployed | 12
Age of CPD(chronic psychotic disorder) onset [Mean (Standard Deviation); unit: years] | 19.89 (4.47)
Duration of CPD(chronic psychotic disorder) [Mean (Standard Deviation); unit: years] | 18.89 (10.87)
Number of previous hospitalizations [Mean (Standard Deviation); unit: hospitalizations]
  For CPD(chronic psychotic disorders) | 6.16 (7.55)
  For substance abuse | 0.05 (0.23)
Past physical abuse [Count of Participants; unit: Participants] | 6
Past sexual abuse [Count of Participants; unit: Participants] | 1
Family history of mental illness [Count of Participants; unit: Participants] | 10
Family history of substance abuse [Count of Participants; unit: Participants] | 10
AUDIT score [Mean (Standard Deviation); unit: units on a scale] — AUDIT: Alcohol Use Disorders Identification Test. There are 10 questions and possible scores range from 0-40. A higher score is associated with worse outcomes for drug/alcohol dependence. Score of 0 suggests abstainer, 1-7 suggests low risk consumption, 8-14 suggests hazardous alcohol consumption, 15+ indicates alcohol dependence.
  units on a scale | 1.84 (3.13)
ASSIST score [Mean (Standard Deviation); unit: units on a scale] — ASSIST: Alcohol, Smoking, and Substance Involvement Screening Test. The ASSIST is an 8 item questionnaire to screen for use of drugs/substances. The ASSIST determines a risk score for each substance. Current frequency of substance use was calculated here using question 2 only. 0-4 was the scale with increasing numbers indicating more drug use frequency. Higher values are associated with worse outcomes/more frequent drug use. 0-3 is lower risk, 4-26 is moderate risk, and 27+ is high risk of dependence to drugs.
  units on a scale | 1.58 (2.65)
Self-reported Charlson Index score [Mean (Standard Deviation); unit: units on a scale] — Self-reported Charlson Index Score. CCI Total Score = the sum of all 10-items, where each item checked gets 1 point, except heart disease and kidney disease which get 2 points each, liver disease which gets 3 points, and cancer and HIV/AIDS which get 6 points each. CCI scores predict risk of mortality. Scores range from 0-24. A higher score is associated with increased risk of mortality.
  units on a scale | 0.37 (0.50)
Body Mass Index(BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.70 (4.89)
Past oral medication history [Count of Participants; unit: Participants]
  Chlorpromazine | 8
  Fluphenizine | 11
  Haloperidol | 14
  Olanzapine | 3
  Promethazine | 8
  Risperidone | 5
Screening TRQ(tablets routine questionnaire) [Mean (Standard Deviation); unit: units on a scale] — Tablets Routine Questionnaire: self-reported proportion of missed oral medication in the last 30 days. Scores range from "0" (perfect adherence) to "100" (did not take any prescribed medication). Mean Tablet Routines Questionnaire calculated only for oral CPD medications (antipsychotics, mood stablizers, antidepressants). If more than 1 oral medication was prescribed. an average TRQ was calculated. Screening sample TRQ, N =19.
  units on a scale | 21.84 (13.83)
Baseline TRQ(tablets routine questionnaire) [Mean (Standard Deviation); unit: units on a scale] — Tablets Routine Questionnaire: self-reported proportion of missed oral medication in the last 30 days. Scores range from "0" (perfect adherence) to "100" (did not take any prescribed medication). Mean Tablet Routines Questionnaire calculated only for oral CPD medications (antipsychotics, mood stablizers, antidepressants). If more than 1 oral medication was prescribed. an average TRQ was calculated. Screening sample TRQ, Baseline sample TRQ, N=18 Population: 18 people were sampled instead of 19 in the baseline.
  units on a scale
    number analyzed (Participants) | 18
    (all) | 12.94 (11.93)

OUTCOME MEASURES:

1. Primary Outcome: Tablets Routine Questionnaire (TRQ)
Description: The TRQ evaluates adherence to medications via a brief self-report instrument that has been validated in populations with bipolar disorder medication adherence. The TRQ identifies nonadherent individuals, defined as those who miss 20-30% or more of their medication in the last week or month. Total scores are represented as a percentage and range from 0 to 100, with higher scores indicating a greater level of nonadherence (higher scores indicate worse adherence to medications).
Time Frame: Change from Baseline to 6 month visit
Population: Since participants stopped using oral medications once they were stable on LAI, there were only two participants remaining at 25 Week visit and therefore analysis was not done. As only 2 individuals were on concommittent oral CPD medication at 25 week follow up, mean change in TRQ was not calculated. This was just done to enter into clinical trials.
Measure: Mean (Standard Deviation); unit: percentage of change in adherence
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 2
percentage of change in adherence
  TRQ Week adherence | -57 (60.8)
  TRQ Month adherence | -23 (0)

2. Primary Outcome: Long-Acting Injectable Adherence (LAI Adherence): Count of Participants Who Received All LAI Injections:
Description: LAI injection adherence will be determined as a count of participants who received LAI injections at the appropriate time (within 7 days of scheduled time).
Time Frame: Baseline to 6 month visit
Population: Poorly adherent patients with schizophrenia who received long-acting injectable antipsychotic medication and a customized adherence enhancement behavioral intervention (CAE-L). LAI injection frequency was 100%.
Measure: Count of Participants; unit: Participants
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Drug Attitude Inventory (DAI)
Description: DAI-10 scoring ranges from -10 to +10 with a total score >0 indicating a positive attitude toward psychiatric medications and a total score of <0 indicating a negative attitude toward psychiatric medications.
Time Frame: Baseline to 6 month visit
Population: Poorly adherent patients with schizophrenia who received long-acting injectable antipsychotic medication and a customized adherence enhancement behavioral intervention (CAE-L).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 18
score on a scale
  Baseline | 7.89 (2.72)
  25 Weeks | 9.83 (0.52)
Statistical Analysis 1: Comparison: CAE + LAI Treatment; Test type: Other — This is a prospective study with a repeated measures design; p = 0.001, t-test, 2 sided — The threshold for statistical significance was p<0.05; It was dependent sample pairwise t-tests, two tailed

4. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: The BPRS measures levels of mania. There are 24 items, scored on a 7-point scale ranging from 0 to 6. Total scores range from 0 to 42, with higher scores indicating higher levels of mania.
Time Frame: Baseline to 6 month visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 18
score on a scale
  Baseline | 27.00 (10.26)
  25-Weeks | 25.06 (8.53)
Statistical Analysis 1: Comparison: CAE + LAI Treatment; Test type: Other — This is a prospective study with a repeated measures design; p = 0.43, t-test, 2 sided — The threshold for statistical significance was p<0.05; It was dependent sample pairwise t-tests, two tailed

5. Secondary Outcome: Clinical Global Impressions (CGI)
Description: The minimum possible score is 1 and the maximum score is 7. A higher score implies a worse condition.
Time Frame: Baseline to 6 month visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 17
units on a scale
  Baseline | 2.88 (1.32)
  25 Weeks | 2.24 (1.09)
Statistical Analysis 1: Comparison: CAE + LAI Treatment; Test type: Other — This is a prospective study with a repeated measures design; p = 0.07, t-test, 2 sided — The threshold for statistical significance was p<0.05; It was dependent sample pairwise t-tests, two tailed

6. Secondary Outcome: Social and Occupational Functioning Scale (SOFAS)
Description: The SOFAS measures social and occupational functioning independent of the overall severity of the individual's psychological symptoms. The minimum score is 0 and the maximum score is 100. A higher rating implies a higher level of functioning.
Time Frame: Baseline to 6 month visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 18
score on a scale
  Baseline | 62.17 (18.28)
  25 Weeks | 68.39 (15.28)
Statistical Analysis 1: Comparison: CAE + LAI Treatment; Test type: Other — This is a prospective study with a repeated measures design; p = 0.10, t-test, 2 sided — The threshold for statistical significance was p<0.05; It was dependent sample pairwise t-tests, two tailed

7. Secondary Outcome: Body Mass Index
Description: Body Mass Index kg/m^2 of participants
Time Frame: Baseline to Month 6(week 25)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 18
kg/m^2
  Baseline | 22.79 (5.02)
  25 Weeks | 22.92 (5.58)
Statistical Analysis 1: Comparison: CAE + LAI Treatment; Test type: Other — This is a prospective study with a repeated measures design; p = 0.75, t-test, 2 sided — The threshold for statistical significance was p<0.05; It was dependent sample pairwise t-tests, two tailed

8. Secondary Outcome: ESRS-A Parkinsonism
Description: Extrapyramidal Symptoms Scale-Abbreviated version for Parkinsonism. It looks at drug-induced Parkinsonism which is made up of motor disturbances. Rigidity, tremor, reduced facial expression/speech, impaired gait/posture, postural instability, and bradykinesia. Each item is rated on a 4 point scale: 0=absent, 3=severe. The higher the value the more severe the Parkinsonism and worst outcomes.
Time Frame: Baseline to 6 months(25 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.06 (0.24)
  25 Weeks | 0.06 (0.24)
Statistical Analysis 1: Comparison: CAE + LAI Treatment; Test type: Other — This is a prospective study with a repeated measures design; p = 1.00, t-test, 2 sided — The threshold for statistical significance was p<0.05; It was dependent sample pairwise t-tests, two tailed

9. Secondary Outcome: ESRS-A Dystonia
Description: Extrapyramidal Symptoms Scale-Abbreviated version for dystonia- drug-induced dystonia is a muscle disorder in which movements are jerky or twisting. Due to the 0.00 values at baseline and 25 weeks, unable to perform t-test and get a p value so no statistical analysis section is reported for this Outcome Measure. Each item is rated on a 4 point scale: 0=absent, 3=severe with the higher numbers indicating worse dystonia and worse outcomes.
Time Frame: Baseline to 6 months(25 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.00 (0.00)
  Week 25 | 0.00 (0.00)

10. Secondary Outcome: ESRS-A Dyskinesia
Description: Extrapyramidal Symptoms Scale-Abbreviated version for Dyskinesia- drug-induced dyskinesia which is repetitive and involuntary movements. Each item is rated on a 4 point scale: 0=absent, 3=severe and higher values indicate greater severity of dyskinesia and worse outcomes.
Time Frame: Baseline to 6 months(25 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.17 (0.51)
  Week 25 | 0.11 (0.47)
Statistical Analysis 1: Comparison: CAE + LAI Treatment; Test type: Other — This is a prospective study with a repeated measures design; p = 0.75, t-test, 2 sided — The threshold for statistical significance was p<0.05; It was dependent sample pairwise t-tests, two tailed

11. Secondary Outcome: ESRS-A Akathisia
Description: Extrapyramidal Symptoms Scale-Abbreviated version for akathisia- drug-induced akathisia consists of inner restlessness and urge to move. Items are measured on a 4 value scale: 0=absent, 3=severe, and higher values indicate more severe akathisia and worse outcomes.
Time Frame: Baseline to 6 months(25 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE + LAI Treatment
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.28 (0.75)
  Week 25 | 0.00 (0.00)
Statistical Analysis 1: Comparison: CAE + LAI Treatment; Test type: Other — This is a prospective study with a repeated measures design; p = 0.14, t-test, 2 sided — The threshold for statistical significance was p<0.05; It was dependent sample pairwise t-tests, two tailed

ADVERSE EVENTS:
Time Frame: 25 weeks
Arm/Group | CAE + LAI Treatment
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 13/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAE + LAI Treatment (N=19)
Substance use relapse and hospitalization (Injury, poisoning and procedural complications) | 1 — 1 participant relapsed into substance abuse and was hospitalized. This SAE was not deemed to be related to individual's participation in the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAE + LAI Treatment (N=19)
Tremor (Nervous system disorders) | 7 — Tremor
Drowsiness (General disorders) | 6 — Drowsiness
Blurry vision (Eye disorders) | 3 — Blurry vision
Restlessness (General disorders) | 2 — Restlessness
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 — Muscle pain

LIMITATIONS AND CAVEATS:
The small sample size, single-site enrollment, and the fact that poor medication adherence was one of the inclusion criterion may make findings less generalizable to the full spectrum of patients with CPD in Tanzania. Additionally, since we did not collect data on family burden, it is not possible to make any conclusions regarding how CAE-L may impact families and communities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT04327843/Prot_SAP_000.pdf
  • Informed Consent Form: Survey ICF UH stamped (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT04327843/ICF_001.pdf
  • Informed Consent Form: English Qualitative Interview (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT04327843/ICF_002.pdf
  • Informed Consent Form: Focus Group ICF (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT04327843/ICF_003.pdf
  • Informed Consent Form: Phase 3 ICF (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT04327843/ICF_004.pdf